CLINICAL TRIAL: NCT01608633
Title: Effects of Spray and Stretch on Postneedling Soreness and Sensitivity After Dry Needling of a Latent Myofascial Trigger Point.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CEU San Pablo University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEU-001
Record Dates: First submitted 2012-05-27; First posted 2012-05-31 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-09

CONDITIONS: Pain After Dry Needling
MeSH Terms: interventions — pentafluoropropane-tetrafluoroethane

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Spray and stretch (Experimental)
  Interventions: Other: Spray and stretch
- Control (No Intervention)

INTERVENTIONS:
Other: Spray and stretch — Physiotherapeutic technique which consist in stretching the muscle while a cold spray is applied on the skin.
  Arms: Spray and stretch

SUMMARY:
Pain after dry needling or injection in the muscle is a frequent secondary effect in the treatment of myofascial pain syndrome. In this trial spray and stretch technique is evaluated as a method to reduce this soreness. As well, the characteristics and the different factors that influence in this pain will be described.

ELIGIBILITY:
Inclusion Criteria:

* Subjects presenting latent trigger points in the trapezius muscle

Exclusion Criteria:

* Subjects with active trigger points or absence of trigger points.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-03; Primary Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Pain | 72 hours
  Visual analogue scale

SECONDARY OUTCOMES:
Pain | 48 hours
  Pressure pain threshold
Psychological factors | 72 hours after needling
  Symptom check list revised. SCL-90-r

CONTACTS AND LOCATIONS:
Locations (1):
- CEU San Pablo University, Madrid, Madrid, Spain